CLINICAL TRIAL: NCT05867992
Title: Proteomic and Metabolomic Detection and Analysis of Serum from Patients with Acute Severe Traumatic Brain Injury: a Prospective, Multicentered Study
Brief Title: Multiomic Analysis of Serum in Acute Period of Traumatic Brain Injury
Acronym: MASTER-TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2024-006
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Biomarker; Multiomic analysis; Diagnosis
MeSH Terms: conditions — Brain Injuries, Traumatic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples from patients with acute severe traumatic brain injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: This group enrolls patients with acute severe traumatic brain injury.
  Interventions: Other: Type of trauma
- Control group: This group enrolls patients with acute traumatic bone fracture but without traumatic brain injury.
  Interventions: Other: Type of trauma

INTERVENTIONS:
Other: Type of trauma — Patients in case group have the severe traumatic brain injury, while patients in control group have the traumatic bone fracture without brain injury.

SUMMARY:
The goal of this experimental observation study is to figure out differently expressed biomarkers in serum in traumatic brain injury patients, compared with bone fracture patients. The main questions it aims to answer are:

1. Which proteins and metabolites are differently expressed in TBI patients' serum?
2. Which proteins or metabolites can serve as the new serum biomarkers for diagnosing TBI? Participants will be treated by routine treatments, and their serum samples will be collected in the emergency room.

DETAILED DESCRIPTION:
This experimental observation study is designed to find out some new characteristics in acute severe traumatic brain injury. To filter the stress response in blood, patients with traumatic fracture are chosen as the control group.

Blood samples of patients who pass the eligibility criteria will be collected immediately in the emergency room. Then the samples will be preprocessed in the laboratory to get serums. These collected serums will be preserved in -80℃ until completing all sample collection. After completing collection, all samples will be sent to proteomic and metabolomic detection. The bioinformatic data will be analyzed to answer these main questions:

1. Which proteins and metabolites are differently expressed in TBI patients' serum? (As a whole characteristic of acute severe TBI)
2. Which proteins or metabolites can serve as the new serum biomarkers for diagnosing TBI? (Deeply digging the value of characteristic of acute severe TBI)

ELIGIBILITY:
Inclusion Criteria:

* With cerebral contusion in 24Hrs for case group, or with traumatic bone fracture in 24Hrs for control group.
* The Glasglow Coma Scale ranges in 3-8 for case group.
* Need to have routine laboratory examination of blood sample.
* Patients or agents sign the informed consent.

Exclusion Criteria:

* With bone fracture for case group, or with brain injury for control group.
* Have Orthopaedic history for case group, or have Neurological history for control group.
* Death in 24 hours.
* Immunosuppressed state.
* Severe multiple organ dysfunction.
* With infection.
* Pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the case group are these with brain injury, caused by trauma and are severe (GCS 3-8) and in acute period (within 12 hours). Meanwhile, these patients should not have acute bone fracture or other orthopaedic diseases, to avoid any biological detecting bias to control group.
  Patients in the control group are these with bone fracture, caused by trauma and in acute period (within 12 hours). Also, these patients should not have acute brain injury or other neurological diseases to avoid the same bias in biological detection.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of differently expressed proteins in patients' serum detected by proteomic | First 12 hours in the emergency room
  Patients' serum will be collected in the emergency room. After collecting all samples, these samples will be detected through proteomic mass spectrometry. The results of proteomic will be further analyzed and compared with control group to filter potential protein biomarkers in serum of severe TBI patients in acute phase.
Number of differently expressed metabolites in patients' serum detected by metabolomic | First 12 hours in the emergency room
  Patients' serum will be collected in the emergency room. After collecting all samples, these samples will be detected through metabolomic mass spectrometry. The results of metabolomic will be further analyzed and compared with control group to filter potential metabolite biomarkers in serum of severe TBI patients in acute phase.

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Feng, Ph.D., Principal Investigator — RenJi Hospital
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided